CLINICAL TRIAL: NCT06413303
Title: The Effect of Experiential Classroom on Establishing Healthy Behaviors During Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: K3955
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Experiential Classroom; Health Behavior; Preconception Education; Adverse Pregnancy Outcome
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiential Classroom Group (Experimental): Participants accept experiential class to establish healthy behaviors. They are also managed continuously through WeChat group chat during prenatal clinical interval.
  Interventions: Behavioral: Experiential Classroom
- Standard Clinic Prenatal Care Group (No Intervention): Participants accept regular routine prenatal care following Chinese standard.

INTERVENTIONS:
Behavioral: Experiential Classroom — Experiential classroom emphasizes putting pregnant women at the center, based on their subjective willingness and previous knowledge and experience, creating an environment for free discussion, exchange, and reflection, and utilizing peer education to fully mobilize the subjective initiative of pregnant women. This approach allows them to explore, discuss, reflect, and learn autonomously, aiming to truly absorb, master, and apply theoretical knowledge.
  Arms: Experiential Classroom Group

SUMMARY:
A multi-center, prospective, randomized controlled clinical trial was conducted to explore the effect of experiential classroom on establishing healthy behaviors during pregnancy.

DETAILED DESCRIPTION:
Adverse pregnancy outcomes, including maternal complications (eg, gestational hypertension, preeclampsia (PE), gestational diabetes mellitus (GDM), placental abruption) and fetal complications (eg, preterm birth, intrauterine growth restriction, large for gestational age (LGA), small for gestational age (SGA), macrosomia) , pose a significant public healthy problem which needs to be addressed. Several studies found that the health status and behaviors of mothers during pregnancy, including dietary patterns, physical activity and emotional well-being, not only affect pregnancy outcomes such as GDM and PE, but also have the long-term implications for the health of the offspring. Therefore, through effective preconception education, helping pregnant women establish healthy behaviors during pregnancy is of great significance in reducing the incidence of adverse pregnancy outcomes. However, traditional educational methods, mostly in the form of face-to-face lectures, have proven to be ineffective. On the other hand, experiential classroom emphasizes putting pregnant women at the center, based on their subjective willingness and previous knowledge and experience, creating an environment for free discussion, exchange, and reflection, and utilizing peer education to fully mobilize the subjective initiative of pregnant women. This approach allows them to explore, discuss, reflect, and learn autonomously, aiming to truly absorb, master, and apply theoretical knowledge. Therefore, to explore the impact of experiential classroom on the establishment of healthy behaviors during pregnancy, we conducted a multicenter, prospective, randomized controlled clinical trial. The study included pregnant women aged 20 and above, married, with singleton pregnancies in early pregnancy, who were randomly assigned to either the experiential classroom group or the routine prenatal care group. Both groups received routine prenatal care. The pregnant women in the personalized exercise guidance group learned about perinatal health knowledge under the guidance of multidisciplinary teachers and were supervised and managed through WeChat groups. The primary outcome measure was the total weight gain during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20.
* Singleton pregnancy.
* The first trimester.
* Be able to undergo regular prenatal follow-ups and delivery in PUMCH.
* Be able to participate in each experiential classroom on time.
* Capable of independently completing questionnaire surveys.

Exclusion Criteria:

* With severe mental illness.
* Severe impairment of liver and kidney function.
* With malignant tumors.
* With contraindications to exercise during pregnancy.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Gestational weight gain | From date of enrollment until the date of delivery.
  Weight before delivery minus weight before pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Liangkun Ma, Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Department of ob gyn, Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No